CLINICAL TRIAL: NCT02494661
Title: Healthy Plate Program in East and South Los Angeles: Testing "Mindfulness-inspired" Video in Community Settings
Brief Title: Nutritional Video Intervention Using Mindfulness-based Principles
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Hortensia Amaro, Dean's Professor, Social Work and Preventive Medicine, Associate Vice Provost, Community Research Initiatives, University of Southern California
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: UP-14-00591
Record Dates: First submitted 2015-06-05; First posted 2015-07-10 (Estimated); Last update posted 2017-03-13 (Actual); Status verified 2017-03

CONDITIONS: Simple Obesity
Keywords: Public Health; Community; Obesity; Hispanic; Women; Nutrition; Mindfulness and stress; Food shopping
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Healthy Cart and Stress Mangement Videos (Experimental): Healthy Cart and Stress Management Videos: Participants receive two nutritional intervention videos: active comparator and managing stress while food shopping.
  Interventions: Behavioral: Healthy Cart and Stress Management Videos
- Healthy Cart Video (Active Comparator): Healthy Cart Video: Participants receive one nutritional video intervention on how to shop for healthy foods using My Plate Guidelines.
  Interventions: Behavioral: Healthy Cart Video

INTERVENTIONS:
Behavioral: Healthy Cart and Stress Management Videos — Healthy Cart and Stress Management Videos: educational videos on healthy food shopping and stress reduction.
  Arms: Healthy Cart and Stress Mangement Videos
Behavioral: Healthy Cart Video — Healthy Cart Video: educational video on healthy food shopping
  Arms: Healthy Cart Video

SUMMARY:
The purpose of this study is to access the acceptability and potential utility of nutritional intervention videos in 1) changing knowledge and attitudes about healthy eating, 2) improving healthy food shopping practices, and 3) enhancing skills for stress reduction during food shopping among low-income Latina mothers.

DETAILED DESCRIPTION:
* Low income Latina mothers (N=218) who are primary grocery shoppers for the family will be recruited through community based organization to take part in the study. Participation will include completion of survey instruments at baseline, immediately following the intervention; and a subset of participants (N=68) will also complete a 2-month follow-up survey and provide up to two weekly grocery store receipts from the prior 1-2 months at baseline and 2-month followup assessment points. The survey will collect data on demographics, knowledge about healthy eating, self efficacy, perceived stress and family history of relevant health issues. Grocery store receipts will be coded and used to evaluate pre-post changes in shopping of healthy vs unhealthy foods. The study compares two conditions: in the control condition, participants will view a 14-minute video on grocery shopping that teaches participants how to make healthy food choices. In the intervention condition, participants will view the aforementioned video in addition to a 15-minute video on how to manage stressors that arise during grocery shopping. -Surveys are to entered manually into chosen database by research assistant.
* 100% of data entries will be checked by Project specialist for accuracy.
* A total of 218 participants will be recruited to partake in the control condition Group A or Group B of the intervention.
* Because of the exploratory nature of the study, power calculations were not used to determine sample size.
* Group x time analyses will compare changes in knowledge, attitudes and self efficacy before and after exposure to the videos in the entire sample; and in the subsample followed for 2 months, compare baseline to 2-month followup changes in knowledge, attitudes, self efficacy, mindfulness and stress related measures as well as behavior change in food choices during grocery shopping.

ELIGIBILITY:
Inclusion Criteria:

* Identify as a Hispanic woman
* Ages: 18-55 years
* Responsible for buying groceries for family
* Language use: Ability to speak, read and write English or Spanish
* Resident in the USC's Health Sciences Campus and University Park Campus neighborhoods

Exclusion Criteria:

* None

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 218 (Actual)
Dates: Start 2014-10; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Change in nutritional knowledge at 2 months | Two months
  All 218 participants will partake in a baseline questionnaire and a post questionnaire immediately following the video intervention to measure knowledge. A subsample of 29 participants from arm A and 39 participants from arm B will also complete a 2-month follow-up questionnaire to measure knowledge at the second time frame.

SECONDARY OUTCOMES:
Change in self-efficacy of healthy food shopping at 2 months | Two months
  All 218 participants will partake in a baseline questionnaire and a post questionnaire immediately following the video intervention to measure knowledge. A subsample of 29 participants from arm A and 39 participants from arm B will also complete a 2-month follow-up questionnaire to measure self-efficacy at the second time frame.
Change in food shopping behavior at 2 months | Two months
  29 participants from arm A and 39 participants from arm B will be asked to turn in 2 grocery store receipts at initial intervention. They will also be asked back for a 2-month follow-up where they will turn in 2 additional receipts to measure changes in grocery shopping behavior.
Change in mindful attention awareness at 2 months | Two months
  29 participants from arm A and 39 participants from arm B will be asked questions regarding mindful attention awareness at initial baseline questionnaire. In addition, they will be asked back for a 2-month follow-up questionnaire to measure changes in mindful attention awareness at the 2-month mark.

CONTACTS AND LOCATIONS:
Overall Officials: Hortensia Amaro, PhD, Principal Investigator — University of Southern California

REFERENCES:
- [Background] Cortes DE, Millan-Ferro A, Schneider K, Vega RR, Caballero AE. Food purchasing selection among low-income, Spanish-speaking Latinos. Am J Prev Med. 2013 Mar;44(3 Suppl 3):S267-73. doi: 10.1016/j.amepre.2012.11.012. PMID 23415192
- [Background] Narayan KM, Boyle JP, Thompson TJ, Sorensen SW, Williamson DF. Lifetime risk for diabetes mellitus in the United States. JAMA. 2003 Oct 8;290(14):1884-90. doi: 10.1001/jama.290.14.1884. PMID 14532317
- [Background] Ogden CL, Carroll MD, Curtin LR, Lamb MM, Flegal KM. Prevalence of high body mass index in US children and adolescents, 2007-2008. JAMA. 2010 Jan 20;303(3):242-9. doi: 10.1001/jama.2009.2012. Epub 2010 Jan 13. PMID 20071470
- [Background] Caballero AE, Bousquet-Santos K, Robles-Osorio L, Montagnani V, Soodini G, Porramatikul S, Hamdy O, Nobrega AC, Horton ES. Overweight Latino children and adolescents have marked endothelial dysfunction and subclinical vascular inflammation in association with excess body fat and insulin resistance. Diabetes Care. 2008 Mar;31(3):576-82. doi: 10.2337/dc07-1540. Epub 2007 Dec 14. PMID 18083792
- [Background] Caballero AE. Type 2 diabetes in the Hispanic or Latino population: challenges and opportunities. Curr Opin Endocrinol Diabetes Obes. 2007 Apr;14(2):151-7. doi: 10.1097/MED.0b013e32809f9531. PMID 17940434
- [Background] Drewnowski A, Darmon N. The economics of obesity: dietary energy density and energy cost. Am J Clin Nutr. 2005 Jul;82(1 Suppl):265S-273S. doi: 10.1093/ajcn/82.1.265S. PMID 16002835
- [Background] Hersey J, Anliker J, Miller C, Mullis RM, Daugherty S, Das S, Bray CR, Dennee P, Sigman-Grant M, Olivia AH. Food shopping practices are associated with dietary quality in low-income households. J Nutr Educ. 2001;33 Suppl 1:S16-26. doi: 10.1016/s1499-4046(06)60066-3. PMID 12857541
- [Background] Powell LM, Chaloupka FJ. Food prices and obesity: evidence and policy implications for taxes and subsidies. Milbank Q. 2009 Mar;87(1):229-57. doi: 10.1111/j.1468-0009.2009.00554.x. PMID 19298422
- [Background] Powell LM, Zhao Z, Wang Y. Food prices and fruit and vegetable consumption among young American adults. Health Place. 2009 Dec;15(4):1064-70. doi: 10.1016/j.healthplace.2009.05.002. Epub 2009 May 14. PMID 19523869
- [Background] Glanz K, Basil M, Maibach E, Goldberg J, Snyder D. Why Americans eat what they do: taste, nutrition, cost, convenience, and weight control concerns as influences on food consumption. J Am Diet Assoc. 1998 Oct;98(10):1118-26. doi: 10.1016/S0002-8223(98)00260-0. PMID 9787717
- [Background] Millan-Ferro A, Caballero AE. Cultural approaches to diabetes self-management programs for the Latino community. Curr Diab Rep. 2007 Oct;7(5):391-7. doi: 10.1007/s11892-007-0064-9. PMID 18173974
- [Background] Malik VS, Fung TT, van Dam RM, Rimm EB, Rosner B, Hu FB. Dietary patterns during adolescence and risk of type 2 diabetes in middle-aged women. Diabetes Care. 2012 Jan;35(1):12-8. doi: 10.2337/dc11-0386. Epub 2011 Nov 10. PMID 22074723
- [Background] Philipson T. The world-wide growth in obesity: an economic research agenda. Health Econ. 2001 Jan;10(1):1-7. doi: 10.1002/1099-1050(200101)10:13.0.co;2-1. No abstract available. PMID 11180565
- [Background] Katz DL, Doughty K, Njike V, Treu JA, Reynolds J, Walker J, Smith E, Katz C. A cost comparison of more and less nutritious food choices in US supermarkets. Public Health Nutr. 2011 Sep;14(9):1693-9. doi: 10.1017/S1368980011000048. Epub 2011 Feb 28. PMID 21356146
- [Background] Perrin JM, Bloom SR, Gortmaker SL. The increase of childhood chronic conditions in the United States. JAMA. 2007 Jun 27;297(24):2755-9. doi: 10.1001/jama.297.24.2755. No abstract available. PMID 17595277
- [Background] Drewnowski A. Obesity and the food environment: dietary energy density and diet costs. Am J Prev Med. 2004 Oct;27(3 Suppl):154-62. doi: 10.1016/j.amepre.2004.06.011. PMID 15450626